CLINICAL TRIAL: NCT00195962
Title: Identification of Risk Factors Among Breast-Fed Infants
Brief Title: Risk Factors of Breastfeeding Study
Status: Completed | Type: Observational
Sponsor: Children's Mercy Hospital Kansas City (Other)
Responsible Party: Susan Teasley, RN, CCRC, Children's Mercy Hospitals and Clinics
Other Study IDs: 040107
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2008-12-18 (Estimated); Status verified 2008-05

CONDITIONS: Healthy
Keywords: Breastfeeding; Post-partum mothers of healthy breast-fed newborns
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

SUMMARY:
The goal of this study is to identify infants who are at risk for developing problems related to being breast-fed.

DETAILED DESCRIPTION:
The goal of this study is to identify infants who are at risk for developing problems related to being breast-fed. A previous study identified items that place an infant at a high risk for developing complications related to being breast-fed. The present study will use the same survey and collect data from more participants. These additional participants are necessary to provide statistical analysis for the survey. The survey being developed will assist health care professionals to identify those infants at risk for developing health problems related to being breast-fed and provide care that will minimize the chances of developing complications.

ELIGIBILITY:
Inclusion Criteria:

* Mothers of healthy infants that are breastfeeding
* At least 24 hours post delivery
* Mother and baby will be dismissed from the hospital together.

Exclusion Criteria:

* Mothers of newborns that are not breastfeeding
* Mothers of newborns that are ill and/or will not be dismissed from the hospital at the same time as the mother

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: * Mothers of healthy infants that are breastfeeding
  * At least 24 hours post delivery
  * Mother and baby will be dismissed from the hospital together.
Sampling Method: Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2004-06; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anne Mercer, RN, Principal Investigator — Children's Mercy Hospital Kansas City
Locations (3):
- United States (3):
  - Children's Mercy Hospitals and Clinics, Kansas City, Missouri
  - Truman Medical Center - Hospital Hill, Kansas City, Missouri
  - Truman Medical Center - Lakewood, Lee's Summit, Missouri

REFERENCES:
- [Background] Hall RT, Mercer AM, Teasley SL, McPherson DM, Simon SD, Santos SR, Meyers BM, Hipsh NE. A breast-feeding assessment score to evaluate the risk for cessation of breast-feeding by 7 to 10 days of age. J Pediatr. 2002 Nov;141(5):659-64. doi: 10.1067/mpd.2002.129081. PMID 12410194